CLINICAL TRIAL: NCT02042248
Title: IGHID 1309 -A Phase I Study to Evaluate the Kinetics of the Immunologic Response and Virologic Impact of AGS-004 in HIV-Infected Individuals Suppressed on Antiretroviral Therapy Initiated During Acute and Chronic HIV Infection
Brief Title: A Phase I Study to Evaluate the Immunologic Response and Virologic Impact of AGS-004
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cynthia L Gay, MD (Other)
Collaborators: Argos Therapeutics (Industry); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Cynthia L Gay, MD, Clinical Assistant Professor, University of North Carolina, Chapel Hill
Organization: University of North Carolina, Chapel Hill (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-3613; DAIDS-ES 11970 (Other: NIH Division of AIDS (DAIDS)); 5U19AI096113-03 (NIH)
Record Dates: First submitted 2014-01-17; First posted 2014-01-22 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: HIV
Keywords: HIV; Acute HIV Infection; Chronic HIV Infection; AGS-004; Phase 1; Antiretroviral Therapy; ART; UNC; Argos Therapeutics; The CARE Collaboratory of AIDS; Immunization; vaccination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: ART initiated during AHI (Experimental): Arm A will enroll approximately 6 participants who initiated ART during AHI (acute HIV infection). The target dose of AGS -004 is delivered in three ID (intradermal) injections of 0.2 mL of AGS-004 (0.6 mL total volume) for a total of 1.2 x 107 viable cells. AGS-004 is administered every 4 weeks at weeks 0, 4, 8, and 12 for a total of 4 doses.
  Interventions: Biological: AGS-004
- Arm B: ART initiated during CHI (Experimental): Arm B will enroll approximately 6 participants who initiated ART during CHI (chronic HIV infection). The target dose of AGS -004 is delivered in three ID (intradermal) injections of 0.2 mL of AGS-004 (0.6 mL total volume) for a total of 1.2 x 107 viable cells. AGS-004 is administered every 4 weeks at weeks 0, 4, 8, and 12 for a total of 4 doses.
  Interventions: Biological: AGS-004

INTERVENTIONS:
Biological: AGS-004 — All participants in both arms will receive the same treatment and doses of AGS-004 in Step 2 at weeks 0, 4, 8, and 12.

SUMMARY:
The purpose of this study is to:

* find out the intensity and duration of the immune response after multiple injections of the investigational study product AGS-004 made from one's own dendritic cells and one's own strain of HIV;
* understand the changes in the body's HIV DNA , and HIV-1 RNA in peripheral and resting CD4+ cells prior to and following administration of AGS- 004.
* find out if low levels of HIV virus that are not detectable by standard HIV RNA assays will decrease following the administration of AGS-004.
* find out if it is safe to give individuals with HIV multiple injections of AGS-004 made from the person's own dendritic cells and their own strain of HIV.
* find out if administration of AGS-004 decreases the amount of latent HIV infection in resting CD4 cells

DETAILED DESCRIPTION:
This is a phase I, single-site, pilot study of the kinetics of the immunological response and virological impact of AGS-004 administered in participants with durable viral suppression on ART initiated during acute (AHI) and chronic HIV infection (CHI). Patients will be screened for eligibility in Step 1. Those meeting study eligibility and with successful production of Argos (AGS)-004 product will then enter Step 2 with administration of AGS-004. All participants will continue ART throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of HIV-1 infection:
* Chronic HIV infection (CHI) is defined as documentation of a positive HIV test result by any licensed ELISA test kit and confirmed by Western blot or Multispot HIV-1/HIV-2 assay prior to screening. HIV culture, HIV antigen, plasma HIV RNA, or a second antibody test by a method other than ELISA is acceptable as an alternative confirmatory test.
* Acute HIV infection (AHI) is defined as a negative or indeterminate enzyme immunoassay (EIA) or a negative HIV RNA test within 45 days of reproducibly detectable plasma HIV RNA by amplification methods.
* Participants in the AHI arm of this study must have initiated ART within 45 days of AHI diagnosis
* Ages ≥ 18 to < 65 years old
* Stable ART regimen for ≥ 6 months prior to Screening (Visit 1) NOTE: The ART regimen is defined by current treatment guidelines. Participants may have had one or more changes in their ART regimen for tolerance, change of guidelines, or dosing simplification.
* On potent antiretroviral therapy, defined as at least 2 nucleoside/nucleotide reverse transcriptase inhibitors plus a non-nucleoside reverse transcriptase inhibitor, integrase inhibitor, or a protease inhibitor. Other potent fully suppressive antiretroviral combinations will be considered on a case-by-case basis. Prior changes in or elimination of medications for easier dosing schedule, intolerance, or toxicity are permitted.
* All participants must continue cART throughout the study.
* Plasma HIV-1 RNA below detected limit by conventional assays (limit of detection determined by assay employed: 75, 50, 40, or 20 copies/mL) for ≥ 1 year
* A single unconfirmed plasma HIV RNA > limit of detection but < 1000 c/mL allowed if a subsequent assay was below the limit of detection; but none in the 6 months preceding the study screening visit.
* Plasma HIV-1 RNA < 50 copies/mL at screening (Visit 1)
* CD4 cell count ≥ 350 cells/mm3 at screening (Visit 1)
* Availability of an adequate sample of frozen plasma (may have been thawed and re-frozen only once) drawn no more than 90 days (and preferably within 30 days) before starting ART, OR an adequate frozen sample of HIV p24 antigen-positive culture supernatant obtained from culture of resting CD4+ T cells.

Note: The VL documented from the pre-ART HIV plasma sample must be ≥8,000 copies/ml before commencing ART regimen (abstracted from medical records). If there is no viral load measurement associated with the pre-ART HIV plasma sample, another pre-ART VL measurement of 8,000 copies/ml can be used to accept the sample for AGS-004 manufacturing.

* No history of auto-immune disease or auto-immune manifestations
* No active HCV infection (measureable HCV RNA) within 90 days of eligibility visit (visit 3).
* No active HBV infection (measureable HBV DNA or HBVsAg+) within 90 days of eligibility visit (visit 3).
* Ability and willingness of participant to give written informed consent
* Able and willing to provide adequate locator information
* Ability and willingness to communicate effectively with study personnel; considered reliable, willing, and cooperative in terms of compliance with the Protocol requirements
* Adequate vascular access for leukapheresis
* Able and willing to receive Intradermal (ID) injections without difficulty
* All female study participants of childbearing potential must agree not to participate in a conception process, and, if participating in sexual activity that could lead to pregnancy, these female participants and their partners must agree to use at least two reliable forms of contraception for at least 21 days prior to study entry and for 12 weeks after the last dose of the study drug product:

  o Acceptable forms of contraception include the following:
* Condoms (male or female) with or without spermicidal agent
* Diaphragm or cervical cap with spermicide
* Intrauterine device (IUD)
* Hormonal birth control drugs given by pills, shots, or placed on or under the skin
* Tubal ligation
* NuvaRing
* Potential participant must have adequate organ function as indicated by the following laboratory values:

System/Laboratory Value:

Hematological:

Absolute neutrophil count (ANC): ≥1,500/mcL Platelets: ≥125,000/mcL Hemoglobin: ≥12g/dL

Coagulation:

Prothrombin Time or INR: ≤1.5x upper limit of normal (ULN)

Chemistry:

K+ levels: Within normal limits Mg++levels: ≥1.2 mEq/L but <1.5 x ULN Glucose: Screening serum glucose (fasting or non-fasting) <120 mg/dl Albumin: ≥3.3 g/dL

Renal:

Serum creatinine or calculated creatinine clearance: ≤1.5 x upper limit of normal (ULN) OR ≥ 60mL/min for potential participants with creatinine levels > 1.3 x institutional ULN

Hepatic:

Serum total bilirubin: Total bilirubin <1.8 times the upper limit of the normal range, unless history of Gilbert's disease or deemed related to treatment with atazanavir. If total bilirubin is elevated, direct bilirubin must be <2 times the ULN range.

AST (SGOT) and ALT (SGPT): ≤ 2.5 X ULN Alkaline Phosphatase: ≤ 2.5 X ULN NOTE: Creatinine clearance should be calculated per institutional standard.

Exclusion Criteria

* HIV-2 antibody positive in the absence of a positive HIV-1 Western Blot as measured at the Screening Visit (Visit 1).
* Untreated syphilis infection (defined as a positive rapid plasma reagin (RPR) without clear documentation of treatment).
* Received any infusion blood product, immune globulin, or hematopoetic growth factors within 90 days prior to study entry.
* History of lymph node irradiation or dissection.
* Use of any of the following within 90 days prior to entry: immunomodulatory, cytokine, or growth stimulating factors such as systemic corticosteroids, cyclosporine, methotrexate, azathioprine, anti-CD25 antibody, IFN, interleukins, interleukin-2 (IL-2), hydroxyurea, thalidomide, sargramostim (granulocyte macrophage-colony stimulating factor [GM-CSF]), dinitrochlorobenzene (DNCB), thymosin alpha, thymopentin, inosiplex, polyribonucleotide, or ditiocarb sodium, coumadin, warfarin, or other Coumadin derivative anticoagulants.
* Use of any prior HIV vaccine (prophylactic and/or therapeutic) within one year before screening (Visit 1).
* Prior participation in AGS-004 clinical research study.
* Treatment interruption of ART for > 1 month since starting the ART from which pre-ART plasma sample was drawn
* For any serious illness requiring systemic treatment or hospitalization, the participant must either complete therapy or be clinically stable on therapy, in the opinion of the site investigator, for at least 90 days prior to entry.
* Pregnancy or breastfeeding
* Any active malignancy that may require chemotherapy or radiation therapy.
* Evidence of hepatic decompensation in cirrhotic participants: history of ascites, hepatic encephalopathy, or bleeding esophageal varices.
* History or other clinical evidence of significant or unstable cardiac disease (e.g., angina, congestive heart failure, recent myocardial infarction, significant arrhythmia) or clinically significant electrocardiogram (ECG) abnormalities. Any history of cardiac rhythm disturbance requiring medical or surgical therapy.
* Any renal disorder deemed clinically significant by the investigator.
* History or other evidence of severe illness, malignancy, immunodeficiency other than HIV, or any other condition that would make the participant unsuitable for the study in the opinion of the investigator.
* Compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric illness or a physical illness, e.g., infectious disease. Prisoner recruitment and participation is not permitted.
* Known allergy or sensitivity to the components of the investigational immunotherapy.
* Use of systemic corticosteroids and use of topical steroids over a total area exceeding 15 cm2 within 30 days prior to Screening or anticipated need for periodic use of corticosteroids during the study.

NOTE: For participants receiving ritonavir (as a booster or protease inhibitor (PI) as part of their ART regimen, the concomitant use of oral/systemic/topical/inhaled/intranasal corticosteroids is prohibited.

* Any history of acute or chronic pancreatitis.
* If the HIV care provider or study investigator is unable, as assessed by the study PI or protocol team, to construct a fully active alternative ART regimen based on previous resistance testing and/or treatment history.
* Known psychiatric or substance abuse disorders that would interfere with one's ability to fully cooperate with the requirements of the trial.
* Any investigational antiretroviral agents or use of a CCR5 inhibitor at Screening.
* Active autoimmune disease or condition including, but not limited to:
* Rheumatoid arthritis (RF positive arthritis with current or recent flare);
* Inflammatory bowel disease;
* Systemic lupus erythematosis (clinical evidence confirmed with ANA >1:80);
* Ankylosing spondylitis; Hashimoto's disease; Scleroderma; Multiple sclerosis; Autoimmune hemolytic anemia (AHA); Immune thrombocytopenic purpura; and, Type I diabetes mellitus (insulin therapy for Type II diabetes is permitted).
* Participation in another investigational clinical research study (with the exception of an antiretroviral treatment trial that uses FDA approved antiretroviral agents) or use of investigational agents within 30 days prior to Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
CD8 T cell responses | 32 weeks
  Measure the duration of HIV-specific CD8 T cell responses by a flow cytometric assay through week 32

SECONDARY OUTCOMES:
Change in low level plasma HIV-1 RNA by single copy assay (SCA) | Weeks 0, 14 and 32
  The change in low level HIV -1 RNA as measured by a single copy assay following AGS-004 administration
Change in frequency of HIV-1 infection of resting CD4+ T cells using the viral outgrowth assay | Weeks 0, 14 and 32
  Change in frequency of HIV-1 infection of resting CD4+ T cells using the viral outgrowth assay following AGS-004 administration

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Gay, MD, MPH, Principal Investigator — University of North Carolina; David Margolis, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finzi D, Hermankova M, Pierson T, Carruth LM, Buck C, Chaisson RE, Quinn TC, Chadwick K, Margolick J, Brookmeyer R, Gallant J, Markowitz M, Ho DD, Richman DD, Siliciano RF. Identification of a reservoir for HIV-1 in patients on highly active antiretroviral therapy. Science. 1997 Nov 14;278(5341):1295-300. doi: 10.1126/science.278.5341.1295. PMID 9360927
- [Background] Finzi D, Blankson J, Siliciano JD, Margolick JB, Chadwick K, Pierson T, Smith K, Lisziewicz J, Lori F, Flexner C, Quinn TC, Chaisson RE, Rosenberg E, Walker B, Gange S, Gallant J, Siliciano RF. Latent infection of CD4+ T cells provides a mechanism for lifelong persistence of HIV-1, even in patients on effective combination therapy. Nat Med. 1999 May;5(5):512-7. doi: 10.1038/8394. PMID 10229227
- [Background] Chun TW, Stuyver L, Mizell SB, Ehler LA, Mican JA, Baseler M, Lloyd AL, Nowak MA, Fauci AS. Presence of an inducible HIV-1 latent reservoir during highly active antiretroviral therapy. Proc Natl Acad Sci U S A. 1997 Nov 25;94(24):13193-7. doi: 10.1073/pnas.94.24.13193. PMID 9371822
- [Background] Schmitz JE, Kuroda MJ, Santra S, Sasseville VG, Simon MA, Lifton MA, Racz P, Tenner-Racz K, Dalesandro M, Scallon BJ, Ghrayeb J, Forman MA, Montefiori DC, Rieber EP, Letvin NL, Reimann KA. Control of viremia in simian immunodeficiency virus infection by CD8+ lymphocytes. Science. 1999 Feb 5;283(5403):857-60. doi: 10.1126/science.283.5403.857. PMID 9933172
- [Background] Addo MM, Draenert R, Rathod A, Verrill CL, Davis BT, Gandhi RT, Robbins GK, Basgoz NO, Stone DR, Cohen DE, Johnston MN, Flynn T, Wurcel AG, Rosenberg ES, Altfeld M, Walker BD. Fully differentiated HIV-1 specific CD8+ T effector cells are more frequently detectable in controlled than in progressive HIV-1 infection. PLoS One. 2007 Mar 28;2(3):e321. doi: 10.1371/journal.pone.0000321. PMID 17389912
- [Background] Goulder PJ, Watkins DI. HIV and SIV CTL escape: implications for vaccine design. Nat Rev Immunol. 2004 Aug;4(8):630-40. doi: 10.1038/nri1417. No abstract available. PMID 15286729
- [Background] Barouch DH, Kunstman J, Kuroda MJ, Schmitz JE, Santra S, Peyerl FW, Krivulka GR, Beaudry K, Lifton MA, Gorgone DA, Montefiori DC, Lewis MG, Wolinsky SM, Letvin NL. Eventual AIDS vaccine failure in a rhesus monkey by viral escape from cytotoxic T lymphocytes. Nature. 2002 Jan 17;415(6869):335-9. doi: 10.1038/415335a. PMID 11797012
- [Background] Vaccari M, Mattapallil J, Song K, Tsai WP, Hryniewicz A, Venzon D, Zanetti M, Reimann KA, Roederer M, Franchini G. Reduced protection from simian immunodeficiency virus SIVmac251 infection afforded by memory CD8+ T cells induced by vaccination during CD4+ T-cell deficiency. J Virol. 2008 Oct;82(19):9629-38. doi: 10.1128/JVI.00893-08. Epub 2008 Jul 30. PMID 18667509
- [Background] McNeil AC, Shupert WL, Iyasere CA, Hallahan CW, Mican JA, Davey RT Jr, Connors M. High-level HIV-1 viremia suppresses viral antigen-specific CD4(+) T cell proliferation. Proc Natl Acad Sci U S A. 2001 Nov 20;98(24):13878-83. doi: 10.1073/pnas.251539598. PMID 11717444
- [Background] Younes SA, Yassine-Diab B, Dumont AR, Boulassel MR, Grossman Z, Routy JP, Sekaly RP. HIV-1 viremia prevents the establishment of interleukin 2-producing HIV-specific memory CD4+ T cells endowed with proliferative capacity. J Exp Med. 2003 Dec 15;198(12):1909-22. doi: 10.1084/jem.20031598. PMID 14676302
- [Background] Lichterfeld M, Yu XG, Mui SK, Williams KL, Trocha A, Brockman MA, Allgaier RL, Waring MT, Koibuchi T, Johnston MN, Cohen D, Allen TM, Rosenberg ES, Walker BD, Altfeld M. Selective depletion of high-avidity human immunodeficiency virus type 1 (HIV-1)-specific CD8+ T cells after early HIV-1 infection. J Virol. 2007 Apr;81(8):4199-214. doi: 10.1128/JVI.01388-06. Epub 2007 Feb 7. PMID 17287271
- [Background] Zanussi S, Simonelli C, D'Andrea M, Caffau C, Clerici M, Tirelli U, DePaoli P. CD8+ lymphocyte phenotype and cytokine production in long-term non-progressor and in progressor patients with HIV-1 infection. Clin Exp Immunol. 1996 Aug;105(2):220-4. doi: 10.1046/j.1365-2249.1996.d01-746.x. PMID 8706325
- [Background] Trautmann L, Janbazian L, Chomont N, Said EA, Gimmig S, Bessette B, Boulassel MR, Delwart E, Sepulveda H, Balderas RS, Routy JP, Haddad EK, Sekaly RP. Upregulation of PD-1 expression on HIV-specific CD8+ T cells leads to reversible immune dysfunction. Nat Med. 2006 Oct;12(10):1198-202. doi: 10.1038/nm1482. Epub 2006 Aug 20. PMID 16917489
- [Background] Steinman RM, Banchereau J. Taking dendritic cells into medicine. Nature. 2007 Sep 27;449(7161):419-26. doi: 10.1038/nature06175. PMID 17898760
- [Background] Nicolette CA, Healey D, Tcherepanova I, Whelton P, Monesmith T, Coombs L, Finke LH, Whiteside T, Miesowicz F. Dendritic cells for active immunotherapy: optimizing design and manufacture in order to develop commercially and clinically viable products. Vaccine. 2007 Sep 27;25 Suppl 2:B47-60. doi: 10.1016/j.vaccine.2007.06.006. Epub 2007 Jun 21. PMID 17669561
- [Background] Osada T, Clay TM, Woo CY, Morse MA, Lyerly HK. Dendritic cell-based immunotherapy. Int Rev Immunol. 2006 Sep-Dec;25(5-6):377-413. doi: 10.1080/08830180600992456. PMID 17169781
- [Background] Connolly NC, Whiteside TL, Wilson C, Kondragunta V, Rinaldo CR, Riddler SA. Therapeutic immunization with human immunodeficiency virus type 1 (HIV-1) peptide-loaded dendritic cells is safe and induces immunogenicity in HIV-1-infected individuals. Clin Vaccine Immunol. 2008 Feb;15(2):284-92. doi: 10.1128/CVI.00221-07. Epub 2007 Oct 17. PMID 17942609
- [Background] Garcia F, Lejeune M, Climent N, Gil C, Alcami J, Morente V, Alos L, Ruiz A, Setoain J, Fumero E, Castro P, Lopez A, Cruceta A, Piera C, Florence E, Pereira A, Libois A, Gonzalez N, Guila M, Caballero M, Lomena F, Joseph J, Miro JM, Pumarola T, Plana M, Gatell JM, Gallart T. Therapeutic immunization with dendritic cells loaded with heat-inactivated autologous HIV-1 in patients with chronic HIV-1 infection. J Infect Dis. 2005 May 15;191(10):1680-5. doi: 10.1086/429340. Epub 2005 Apr 11. PMID 15838795
- [Background] Lu W, Arraes LC, Ferreira WT, Andrieu JM. Therapeutic dendritic-cell vaccine for chronic HIV-1 infection. Nat Med. 2004 Dec;10(12):1359-65. doi: 10.1038/nm1147. Epub 2004 Nov 28. PMID 15568033
- [Background] Whiteside TL, Piazza P, Reiter A, Stanson J, Connolly NC, Rinaldo CR Jr, Riddler SA. Production of a dendritic cell-based vaccine containing inactivated autologous virus for therapy of patients with chronic human immunodeficiency virus type 1 infection. Clin Vaccine Immunol. 2009 Feb;16(2):233-40. doi: 10.1128/CVI.00066-08. Epub 2008 Nov 26. PMID 19038780
- [Background] Ide F, Nakamura T, Tomizawa M, Kawana-Tachikawa A, Odawara T, Hosoya N, Iwamoto A. Peptide-loaded dendritic-cell vaccination followed by treatment interruption for chronic HIV-1 infection: a phase 1 trial. J Med Virol. 2006 Jun;78(6):711-8. doi: 10.1002/jmv.20612. PMID 16628588
- [Background] Maldarelli F, Palmer S, King MS, Wiegand A, Polis MA, Mican J, Kovacs JA, Davey RT, Rock-Kress D, Dewar R, Liu S, Metcalf JA, Rehm C, Brun SC, Hanna GJ, Kempf DJ, Coffin JM, Mellors JW. ART suppresses plasma HIV-1 RNA to a stable set point predicted by pretherapy viremia. PLoS Pathog. 2007 Apr;3(4):e46. doi: 10.1371/journal.ppat.0030046. PMID 17411338
- [Background] Palmer S, Maldarelli F, Wiegand A, Bernstein B, Hanna GJ, Brun SC, Kempf DJ, Mellors JW, Coffin JM, King MS. Low-level viremia persists for at least 7 years in patients on suppressive antiretroviral therapy. Proc Natl Acad Sci U S A. 2008 Mar 11;105(10):3879-84. doi: 10.1073/pnas.0800050105. Epub 2008 Mar 10. PMID 18332425
- [Background] Archin NM, Liberty AL, Kashuba AD, Choudhary SK, Kuruc JD, Crooks AM, Parker DC, Anderson EM, Kearney MF, Strain MC, Richman DD, Hudgens MG, Bosch RJ, Coffin JM, Eron JJ, Hazuda DJ, Margolis DM. Administration of vorinostat disrupts HIV-1 latency in patients on antiretroviral therapy. Nature. 2012 Jul 25;487(7408):482-5. doi: 10.1038/nature11286. PMID 22837004
- [Background] Shan L, Deng K, Shroff NS, Durand CM, Rabi SA, Yang HC, Zhang H, Margolick JB, Blankson JN, Siliciano RF. Stimulation of HIV-1-specific cytolytic T lymphocytes facilitates elimination of latent viral reservoir after virus reactivation. Immunity. 2012 Mar 23;36(3):491-501. doi: 10.1016/j.immuni.2012.01.014. Epub 2012 Mar 8. PMID 22406268
- [Background] DeBenedette MA, Calderhead DM, Ketteringham H, Gamble AH, Horvatinovich JM, Tcherepanova IY, Nicolette CA, Healey DG. Priming of a novel subset of CD28+ rapidly expanding high-avidity effector memory CTL by post maturation electroporation-CD40L dendritic cells is IL-12 dependent. J Immunol. 2008 Oct 15;181(8):5296-305. doi: 10.4049/jimmunol.181.8.5296. PMID 18832685
- [Background] Calderhead DM, DeBenedette MA, Ketteringham H, Gamble AH, Horvatinovich JM, Tcherepanova IY, Nicolette CA, Healey DG. Cytokine maturation followed by CD40L mRNA electroporation results in a clinically relevant dendritic cell product capable of inducing a potent proinflammatory CTL response. J Immunother. 2008 Oct;31(8):731-41. doi: 10.1097/CJI.0b013e318183db02. PMID 18779746
- [Background] Tcherepanova I, Harris J, Starr A, Cleveland J, Ketteringham H, Calderhead D, Horvatinovich J, Healey D, Nicolette CA. Multiplex RT-PCR amplification of HIV genes to create a completely autologous DC-based immunotherapy for the treatment of HIV infection. PLoS One. 2008 Jan 30;3(1):e1489. doi: 10.1371/journal.pone.0001489. PMID 18231576
- [Background] Addo MM, Yu XG, Rosenberg ES, Walker BD, Altfeld M. Cytotoxic T-lymphocyte (CTL) responses directed against regulatory and accessory proteins in HIV-1 infection. DNA Cell Biol. 2002 Sep;21(9):671-8. doi: 10.1089/104454902760330219. PMID 12396610
- [Background] Van Gulck ER, Ponsaerts P, Heyndrickx L, Vereecken K, Moerman F, De Roo A, Colebunders R, Van den Bosch G, Van Bockstaele DR, Van Tendeloo VF, Allard S, Verrier B, Maranon C, Hoeffel G, Hosmalin A, Berneman ZN, Vanham G. Efficient stimulation of HIV-1-specific T cells using dendritic cells electroporated with mRNA encoding autologous HIV-1 Gag and Env proteins. Blood. 2006 Mar 1;107(5):1818-27. doi: 10.1182/blood-2005-01-0339. Epub 2005 Nov 1. PMID 16263796
- [Background] Altfeld M, Addo MM, Eldridge RL, Yu XG, Thomas S, Khatri A, Strick D, Phillips MN, Cohen GB, Islam SA, Kalams SA, Brander C, Goulder PJ, Rosenberg ES, Walker BD; HIV Study Collaboration. Vpr is preferentially targeted by CTL during HIV-1 infection. J Immunol. 2001 Sep 1;167(5):2743-52. doi: 10.4049/jimmunol.167.5.2743. PMID 11509618
- [Background] Novitsky V, Cao H, Rybak N, Gilbert P, McLane MF, Gaolekwe S, Peter T, Thior I, Ndung'u T, Marlink R, Lee TH, Essex M. Magnitude and frequency of cytotoxic T-lymphocyte responses: identification of immunodominant regions of human immunodeficiency virus type 1 subtype C. J Virol. 2002 Oct;76(20):10155-68. doi: 10.1128/jvi.76.20.10155-10168.2002. PMID 12239290
- [Background] Quaranta MG, Mattioli B, Giordani L, Viora M. The immunoregulatory effects of HIV-1 Nef on dendritic cells and the pathogenesis of AIDS. FASEB J. 2006 Nov;20(13):2198-208. doi: 10.1096/fj.06-6260rev. PMID 17077296
- [Background] Majumder B, Janket ML, Schafer EA, Schaubert K, Huang XL, Kan-Mitchell J, Rinaldo CR Jr, Ayyavoo V. Human immunodeficiency virus type 1 Vpr impairs dendritic cell maturation and T-cell activation: implications for viral immune escape. J Virol. 2005 Jul;79(13):7990-8003. doi: 10.1128/JVI.79.13.7990-8003.2005. PMID 15956545
- [Background] Tcherepanova I, Starr A, Lackford B, Adams MD, Routy JP, Boulassel MR, Calderhead D, Healey D, Nicolette C. The immunosuppressive properties of the HIV Vpr protein are linked to a single highly conserved residue, R90. PLoS One. 2009 Jun 10;4(6):e5853. doi: 10.1371/journal.pone.0005853. PMID 19516896
- [Background] Morse MA, Coleman RE, Akabani G, Niehaus N, Coleman D, Lyerly HK. Migration of human dendritic cells after injection in patients with metastatic malignancies. Cancer Res. 1999 Jan 1;59(1):56-8. PMID 9892184
- [Background] Serody JS, Collins EJ, Tisch RM, Kuhns JJ, Frelinger JA. T cell activity after dendritic cell vaccination is dependent on both the type of antigen and the mode of delivery. J Immunol. 2000 May 1;164(9):4961-7. doi: 10.4049/jimmunol.164.9.4961. PMID 10779807
- [Background] Routy JP, Boulassel MR, Yassine-Diab B, Nicolette C, Healey D, Jain R, Landry C, Yegorov O, Tcherepanova I, Monesmith T, Finke L, Sekaly RP. Immunologic activity and safety of autologous HIV RNA-electroporated dendritic cells in HIV-1 infected patients receiving antiretroviral therapy. Clin Immunol. 2010 Feb;134(2):140-7. doi: 10.1016/j.clim.2009.09.009. Epub 2009 Nov 4. PMID 19889582
- [Background] Rosenberg ES, Billingsley JM, Caliendo AM, Boswell SL, Sax PE, Kalams SA, Walker BD. Vigorous HIV-1-specific CD4+ T cell responses associated with control of viremia. Science. 1997 Nov 21;278(5342):1447-50. doi: 10.1126/science.278.5342.1447. PMID 9367954
- [Background] Rosenberg ES, Altfeld M, Poon SH, Phillips MN, Wilkes BM, Eldridge RL, Robbins GK, D'Aquila RT, Goulder PJ, Walker BD. Immune control of HIV-1 after early treatment of acute infection. Nature. 2000 Sep 28;407(6803):523-6. doi: 10.1038/35035103. PMID 11029005
- [Background] Volberding P, Demeter L, Bosch RJ, Aga E, Pettinelli C, Hirsch M, Vogler M, Martinez A, Little S, Connick E; ACTG 371 Team. Antiretroviral therapy in acute and recent HIV infection: a prospective multicenter stratified trial of intentionally interrupted treatment. AIDS. 2009 Sep 24;23(15):1987-95. doi: 10.1097/QAD.0b013e32832eb285. PMID 19696651
- [Background] Hecht FM, Wang L, Collier A, Little S, Markowitz M, Margolick J, Kilby JM, Daar E, Conway B, Holte S; AIEDRP Network. A multicenter observational study of the potential benefits of initiating combination antiretroviral therapy during acute HIV infection. J Infect Dis. 2006 Sep 15;194(6):725-33. doi: 10.1086/506616. Epub 2006 Aug 15. PMID 16941337
- [Background] Ortiz GM, Nixon DF, Trkola A, Binley J, Jin X, Bonhoeffer S, Kuebler PJ, Donahoe SM, Demoitie MA, Kakimoto WM, Ketas T, Clas B, Heymann JJ, Zhang L, Cao Y, Hurley A, Moore JP, Ho DD, Markowitz M. HIV-1-specific immune responses in subjects who temporarily contain virus replication after discontinuation of highly active antiretroviral therapy. J Clin Invest. 1999 Sep;104(6):R13-8. doi: 10.1172/JCI7371. PMID 10491418
- [Background] Bongiovanni M, Casana M, Tincati C, d'Arminio Monforte A. Treatment interruptions in HIV-infected subjects. J Antimicrob Chemother. 2006 Sep;58(3):502-5. doi: 10.1093/jac/dkl268. Epub 2006 Jul 1. PMID 16816398
- [Background] Rosenberg ZF, Fauci AS. Immunopathogenic mechanisms of HIV infection: cytokine induction of HIV expression. Immunol Today. 1990 May;11(5):176-80. doi: 10.1016/0167-5699(90)90070-p. PMID 2186752
- [Background] Pilcher CD, Eron JJ Jr, Galvin S, Gay C, Cohen MS. Acute HIV revisited: new opportunities for treatment and prevention. J Clin Invest. 2004 Apr;113(7):937-45. doi: 10.1172/JCI21540. PMID 15057296
- [Background] Pires A, Hardy G, Gazzard B, Gotch F, Imami N. Initiation of antiretroviral therapy during recent HIV-1 infection results in lower residual viral reservoirs. J Acquir Immune Defic Syndr. 2004 Jul 1;36(3):783-90. doi: 10.1097/00126334-200407010-00004. PMID 15213561
- [Background] Ramratnam B, Ribeiro R, He T, Chung C, Simon V, Vanderhoeven J, Hurley A, Zhang L, Perelson AS, Ho DD, Markowitz M. Intensification of antiretroviral therapy accelerates the decay of the HIV-1 latent reservoir and decreases, but does not eliminate, ongoing virus replication. J Acquir Immune Defic Syndr. 2004 Jan 1;35(1):33-7. doi: 10.1097/00126334-200401010-00004. PMID 14707789
- [Background] Chamberland A, Sylla M, Boulassel MR, Baril JG, Cote P, Thomas R, Trottier B, Rouleau D, Routy JP, Tremblay C; Investigators of the Primary HIV-Infection Cohort of Montreal. Effect of antiretroviral therapy on HIV-1 genetic evolution during acute infection. Int J STD AIDS. 2011 Mar;22(3):146-50. doi: 10.1258/ijsa.2010.010292. PMID 21464451
- [Background] Keedy KS, Archin NM, Gates AT, Espeseth A, Hazuda DJ, Margolis DM. A limited group of class I histone deacetylases acts to repress human immunodeficiency virus type 1 expression. J Virol. 2009 May;83(10):4749-56. doi: 10.1128/JVI.02585-08. Epub 2009 Mar 11. PMID 19279091
- [Background] Yukl SA, Boritz E, Busch M, Bentsen C, Chun TW, Douek D, Eisele E, Haase A, Ho YC, Hutter G, Justement JS, Keating S, Lee TH, Li P, Murray D, Palmer S, Pilcher C, Pillai S, Price RW, Rothenberger M, Schacker T, Siliciano J, Siliciano R, Sinclair E, Strain M, Wong J, Richman D, Deeks SG. Challenges in detecting HIV persistence during potentially curative interventions: a study of the Berlin patient. PLoS Pathog. 2013;9(5):e1003347. doi: 10.1371/journal.ppat.1003347. Epub 2013 May 9. PMID 23671416
- [Background] Azzoni L, Foulkes AS, Papasavvas E, Mexas AM, Lynn KM, Mounzer K, Tebas P, Jacobson JM, Frank I, Busch MP, Deeks SG, Carrington M, O'Doherty U, Kostman J, Montaner LJ. Pegylated Interferon alfa-2a monotherapy results in suppression of HIV type 1 replication and decreased cell-associated HIV DNA integration. J Infect Dis. 2013 Jan 15;207(2):213-22. doi: 10.1093/infdis/jis663. Epub 2012 Oct 26. PMID 23105144
- [Background] Liszewski MK, Yu JJ, O'Doherty U. Detecting HIV-1 integration by repetitive-sampling Alu-gag PCR. Methods. 2009 Apr;47(4):254-60. doi: 10.1016/j.ymeth.2009.01.002. Epub 2009 Feb 3. PMID 19195495
- [Background] Palmer S, Wiegand AP, Maldarelli F, Bazmi H, Mican JM, Polis M, Dewar RL, Planta A, Liu S, Metcalf JA, Mellors JW, Coffin JM. New real-time reverse transcriptase-initiated PCR assay with single-copy sensitivity for human immunodeficiency virus type 1 RNA in plasma. J Clin Microbiol. 2003 Oct;41(10):4531-6. doi: 10.1128/JCM.41.10.4531-4536.2003. PMID 14532178
- [Background] Archin NM, Eron JJ, Palmer S, Hartmann-Duff A, Martinson JA, Wiegand A, Bandarenko N, Schmitz JL, Bosch RJ, Landay AL, Coffin JM, Margolis DM. Valproic acid without intensified antiviral therapy has limited impact on persistent HIV infection of resting CD4+ T cells. AIDS. 2008 Jun 19;22(10):1131-5. doi: 10.1097/QAD.0b013e3282fd6df4. PMID 18525258
- [Background] Gandhi RT, Zheng L, Bosch RJ, Chan ES, Margolis DM, Read S, Kallungal B, Palmer S, Medvik K, Lederman MM, Alatrakchi N, Jacobson JM, Wiegand A, Kearney M, Coffin JM, Mellors JW, Eron JJ; AIDS Clinical Trials Group A5244 team. The effect of raltegravir intensification on low-level residual viremia in HIV-infected patients on antiretroviral therapy: a randomized controlled trial. PLoS Med. 2010 Aug 10;7(8):e1000321. doi: 10.1371/journal.pmed.1000321. PMID 20711481
- [Background] Tcherepanova, I, Harri, J, Horvatinovich, J, et al. Autologous dendritic cell based therapy modulates proviral DNA levels in chronically HIV-infected subjects. AIDS Vaccine 2013 7 - 10 October in Barcelona, Spain.
- [Background] Wolf J, Bogner C, Hoffmann V, Avettand-Fenoel K, Schewe R, Pauli J, et al. 5-drug HAART during primary HIV infection leads to a reduction of proviral DNA levels in comparison to levels achievable during chronic infection. In: 7th IAS Conference on HIV Pathogenesis. Kuala Lumpur, Malaysia; 2013.
- See also: University of North Carolina website — http://www.unc.edu